CLINICAL TRIAL: NCT07010718
Title: Comparative Effectiveness Trial of Sleep Promotion vs. Disruption in High Suicide Risk Inpatients
Brief Title: Improving Sleep in a Psychiatric Hospital
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Michelle Patriquin, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HSC-MS-24-1035
Record Dates: First submitted 2025-05-23; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Sleep Disorder; Mental Health Issue
Keywords: suicidal ideation
MeSH Terms: conditions — Sleep Wake Disorders; Suicidal Ideation | interventions — Odorants; Ear Protective Devices

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sleep promotion (Experimental): Scented Oil Ear Plugs Eye Mask Video based safety checks will be done as long as participant is asleep. In person safety check will be done once participant is awake
  Interventions: Drug: Scented Oil; Device: Ear Plugs; Device: Eye Mask; Behavioral: Video based safety check; Behavioral: In person safety check
- Treatment as usual (Active Comparator): Only in person safety check will be conducted
  Interventions: Behavioral: In person safety check

INTERVENTIONS:
Drug: Scented Oil — inpatient-safe aromatherapy (scented oil)
  Arms: Sleep promotion
Device: Ear Plugs — ingestible-safe ear plugs (noise blocking)
  Arms: Sleep promotion
Device: Eye Mask — inpatient-safe eye mask (light blocking).
  Arms: Sleep promotion
Behavioral: Video based safety check — video based safety checks will be conducted as long as participants are in bed and asleep
  Arms: Sleep promotion
Behavioral: In person safety check — In person safety checks will be conducted every 30 minutes

SUMMARY:
The purpose of this study is to examine effects of sleep promotion versus treatment as usual (TAU) on subjective, self-reported sleep while in inpatient psychiatric treatment, to examine effects of sleep promotion vs. TAU/sleep disruption on self-reported depression, anxiety, suicide risk across inpatient length of stay, readmission at 72 hours, objective sleep and to compare implementation outcomes of acceptability and feasibility of sleep promotion relative to TAU/sleep disruption as reported by patients, clinicians, and clinic leaders using mixed methods.

ELIGIBILITY:
Inclusion Criteria:

* Admitted voluntarily to inpatient psychiatric hospital for suicidal ideation or behavior.
* Continue to express suicide risk on the Suicide Behaviors Questionnaire-Revised (SBQ-R) of ≥8 at admission.
* Cognitive ability as tested by the Montreal Cognitive Assessment (MoCA) of > 23.
* Have sufficient communication and comprehension ability to consent to the study
* English speaking

Exclusion Criteria:

* Intellectual disability/unable to give informed consent.
* Patients with one-to-one supervision or 15-minute (Q15) safety checks for suicidality or aggression will be unable to enroll in the study until these restrictions are discontinued.
* Patients with roommates that are on one-to-one supervision or Q15 safety checks for suicidality or aggression.
* Patients enrolled in the study with a patient admitted as their roommate who requires one-to-one supervision or Q15 checks-Patient will be unenrolled if a room change is not possible.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in nighttime Sleep Quality as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Admission, Discharge (about 2 weeks after admission )
  The PSQI has 19 self rated questions with a global score range of 0 to 21.It has 7 components and each is scored from 0 (no difficulty) to 3(severe difficulty) with higher scores indicating poorer sleep quality.
Change in insomnia as assessed by the Insomnia Severity Index (ISI) | Admission, Discharge (about 2 weeks after admission )
  The ISI is a 7-item , each item is rated on a 0 (no problem)-4 (very severe problem) scale, with total scores ranging from 0 to 28. Higher scores indicate greater insomnia severity.
Change in daytime Sleepiness as assessed by the Epworth Sleepiness Scale (ESS) | Admission, Discharge (about 2 weeks after admission )
  The ESS is an 8-item questionnaire. Each item is scored from 0 (would never doze) to 3 (high chance of dozing). The total score ranges from 0 to 24, with higher scores indicating greater daytime sleepiness.

SECONDARY OUTCOMES:
Change in suicide risk as assessed by the Suicide Behaviors Questionnaire Revised (SBQ-R) | Admission, Discharge (about 2 weeks after admission )
  The SBQ-R is a 4-item questionnaire, each scored on a different scale. Total scores range from 3 to 18, with higher scores indicating greater suicide risk.
  Item 1 is scored from 1 [Never (1 point)] to 6 [I have attempted to kill myself more than once (6 points)] Item2 is scored from 1[Never (1 point)] to 5[Very often (5 or more times) (5 points)] Item 3 is scored from 1[No (1 point)] to 5[Yes, more than once, and really wanted to do it (5 points)] Item 3 is scored from 1[Never (1 point)] to 6 [Rather likely (6 points)]
Change in Suicide Ideation as assessed by the Beck Scale for Suicide Ideation (BSS) | Admission, Discharge (about 2 weeks after admission )
  The Beck Scale for Suicide Ideation (BSS) is a 21-item questionnaire. The first 19 items are scored from 0(No ideation/symptom) to 2 (Severe ideation/symptom) for a maximum score of 38, higher scores indicate greater severity of suicidal ideation.
  The last 2 items assess past suicide attempts and intent to die during the most recent attempt. These are not included in the total score.
Change in Anxiety as assessed by the Generalized Anxiety Disorder (GAD-7) scale | Admission, Discharge (about 2 weeks after admission )
  The GAD-7 is a brief, 7-item questionnaire, and each is scored from 0(not at all) to 3( nearly every day) for a total score range of 0-21, higher score indicating severe anxiety symptoms
Change in Depression as assessed by the Patient Health Questionnaire (PHQ-9) | Admission, Discharge (about 2 weeks after admission )
  The PHQ-9 is a 9-item questionnaire, each is scored from 0( not at all) to 3(nearly every day) for a total score range of 0-27, higher scores indicate greater severity of depressive symptoms.
Objective Nighttime Sleep Quantity as assessed by the Total Sleep Time (TST) via ActiGraph wGT3X-BT | Each night during length of stay (about 2 weeks)
  Total Sleep Time (TST) is the total amount of actual sleep time recorded during the nighttime sleep period. This measure is objectively assessed using the ActiGraph wGT3X-BT, a validated wrist-worn accelerometer device that estimates sleep parameters based on movement data.TST is calculated as the sum of all sleep epochs during the main sleep period (typically nighttime) and is reported in minutes or hours.
Objective Nighttime Sleep Quality as assessed by the Nighttime Awakenings via ActiGraph wGT3X-BT | Each night during length of stay(about 2 weeks)
  Nighttime Awakenings refer to the number and/or duration of awakenings during the main sleep period, objectively measured by the ActiGraph wGT3X-BT wrist-worn accelerometer. The device detects movement patterns to identify sleep interruptions, providing an estimate of sleep fragmentation and overall sleep quality.
  The outcome will be reported as: Total number of awakenings per night

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Patriquin, PhD, ABPP, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No